CLINICAL TRIAL: NCT04834973
Title: A Phase Ib/IIa, Dose-escalation Study to Evaluate the Safety, Tolerability, and Preliminary Effectiveness of Intratumoural Tigilanol Tiglate in Combination With Intravenous Pembrolizumab in Adults With Stage IIIb to IV M1c-melanoma
Brief Title: A Trial of Tigilanol Tiglate in Combination With Pembrolizumab in Stage IIIB to IV M1c-melanoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Insufficient Patient Recruitment Rates
Sponsor: QBiotics Group Limited (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QB46C-H06; KN-B16 (Other: Merck); U1111-1258-4085 (Other: WHO Universal Trial Number (UTN))
Record Dates: First submitted 2021-03-29; First posted 2021-04-08 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Melanoma
Keywords: Melanoma; Intratumoural; Tigilanol Tiglate; Pembrolizumab; Keytruda; Epoxytigilane
MeSH Terms: conditions — Melanoma | interventions — EBC-46; pembrolizumab

STUDY DESIGN:
Intervention Model Description: Standard 3 + 3 Dose escalation study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single arm open label (Experimental): Single or multiple Intratumoural treatment of tigilanol tiglate at escalating doses of 0.6 mg/m2, 1.2 mg/m2 and 2.4 mg/m2 given every 28 days (+1 to 14days) in combination with three weekly 200 mg intravenous doses of pembrolizumab.
  Interventions: Drug: tigilanol tiglate; Drug: pembrolizumab

INTERVENTIONS:
Drug: tigilanol tiglate — Single or multiple Intratumoural treatment of tigilanol tiglate at escalating doses of 0.6 mg/m2, 1.2 mg/m2 and 2.4 mg/m2.
  Tigilanol tiglate is a novel, short-chain diterpene ester in early clinical development for local treatment of a wide range of solid tumours.
  Other Names: EBC-46
Drug: pembrolizumab — Three weekly 200 mg intravenous pembrolizumab treatment.
  Pembrolizumab is a systemic anti-programmed cell death receptor 1 (PD 1) immunotherapy.
  Other Names: Keytruda

SUMMARY:
A Phase Ib/IIa, multicentre, open label, dose-escalation study to evaluate the safety, tolerability, and preliminary effectiveness of intratumoural tigilanol tiglate in combination with intravenous pembrolizumab in adult patients with unresectable, Stage IIIB to IV M1c melanoma.

DETAILED DESCRIPTION:
Intratumoural treatment with tigilanol tiglate combined with systemic anti-programmed cell death receptor 1 (PD 1) immunotherapy may enhance anti-tumour immune responses and improve outcomes for patients with melanoma.

Primary Objectives:

1. To determine the maximum tolerated dose (MTD) or maximum feasible dose (MFD) level of a single intratumoural treatment of tigilanol tiglate (Tx1) administered in combination with pembrolizumab.

2. To assess the safety and tolerability of: i) A single treatment (Tx1) of intratumoural tigilanol tiglate at escalating dose levels (dose-escalation) administered in combination with intravenous (IV) pembrolizumab (200 mg); and ii) Repeat treatments of intratumoural tigilanol tiglate (maximum of 3 treatments) administered in combination with IV pembrolizumab (200 mg, Q3W). Repeat treatment(s) of intratumoural tigilanol tiglate to be administered at the same dose level at Tx1 as follows:

1. If the initially injected tumour(s) are not fully ablated, then intratumoural tigilanol tiglate Tx2 +/- Tx3 may be re-administered to the same tumour(s).
2. If the initially injected tumour(s) are fully ablated and additional pre-identified tumours can be treated, then intratumoural tigilanol tiglate, Tx2 +/- Tx3 may also be administered to those tumours.

Note: Tumours identified at Screening that are designated as "not to be injected" tumours (i.e. non-injected tumours for observation) cannot be treated at Tx1, Tx2 or Tx3.

Secondary Objectives:

1. To evaluate tumour response according to RECIST 1.1 criteria, including loco-regional control of injected tumour(s) and non-injected tumour(s), and survival in patients treated in this study.
2. To assess the safety and tolerability of ongoing treatment with pembrolizumab up to a total of 35 cycles (Q3W), including the combination with up to 3 treatments of intratumoural tigilanol tiglate (Q3W).

Exploratory Objectives:

1. To evaluate the tumour response of tumours following treatment with intratumoural injection with tigilanol tiglate in combination with pembrolizumab

ELIGIBILITY:
Inclusion Criteria:

A patient will be eligible for study participation if they meet ALL of the following criteria:

1. Are willing and able to provide written informed consent for the study prior to any protocol-required procedures and to comply with all local and study requirements. (Note: If a patient is unable to provide written informed consent, a legally acceptable representative may provide consent on their behalf).
2. Are an adult at least 18 years of age on the day of providing informed consent.
3. Have a histologically confirmed diagnosis of melanoma that is Stage IIIB to IV M1c (AJCC 8th Ed.) for whom surgery is not recommended. Only patients previously exposed to a checkpoint inhibitor are eligible. Prior BRAF inhibitor therapy is allowed for BRAF V600+ patients.
4. Have measurable disease per RECIST v1.1 including cutaneous or subcutaneous tumours, or regional lymph nodes consisting of ≥ 1 target tumour accessible and amenable to intratumoural injection and ≥ 1 target tumour designated as a non-injected tumour for observation that can be accurately measured by contrast enhanced CT or MRI as assessed by the Investigator's local site radiology.
5. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
6. Have life expectancy of more than 12 weeks.
7. Have adequate organ function as defined below. Specimens must be collected within 10 days prior to the start of study treatment.

   Haematological:

   Absolute neutrophil count (ANC) ≥ 1500/µL Platelets ≥ 100 000/µL Haemoglobin ≥ 9.0 g/dL OR ≥ 5.6 mmol/L1

   Renal

   Creatinine OR Measured or calculated2 creatinine clearance (GFR can also be used in place of creatinine or CrCl) ≤ 1.5 × ULN OR

   ≥ 30 mL/min for patient with creatinine levels > 1.5 × institutional ULN

   Hepatic

   Total bilirubin: ≤ 1.5 × ULN OR direct bilirubin ≤ ULN for patients with total bilirubin levels > 1.5 × ULN

   AST (SGOT) and ALT (SGPT) ≤ 2.5 × ULN (≤ 5 × ULN for patients with liver metastases)

   Coagulation

   International normalized ratio (INR) OR prothrombin time (PT) Activated partial thromboplastin time (aPTT): ≤ 1.5 × ULN unless patient is receiving anticoagulant therapy as long as PT or aPTT is within therapeutic range of intended use of anticoagulants
8. Meet the following conditions:

   1. A male patient must agree to use adequate contraception (as defined below) from the first day of Screening prior to study entry, for the duration of study participation, and for at least 90 days (one spermatogenesis cycle) following their last treatment day. Additionally, male patients must agree to not donate sperm or father children for the duration of study participation and for at least 90 days following their last treatment day.
   2. A female patient is eligible to participate if she is not pregnant (as demonstrated by negative serum beta-human chorionic gonadotropin [βhCG] pregnancy test), not breastfeeding, agrees to not conceive children for at least 120 days following their last study treatment day, and at least one of the following conditions applies:

   i) Not a woman of childbearing potential (WOCBP) (i.e., pre-menarchal, surgically permanently sterile [hysterectomy, bilateral salpingectomy and bilateral oophorectomy] or ≥ 12 months post-menopausal without an alternative medical cause), or

ii) A WOCBP (i.e., not pre-menarchal, not surgically permanently sterile [hysterectomy, bilateral salpingectomy and bilateral oophorectomy] or not ≥ 12 months post-menopausal without an alternative medical cause), who agrees to use adequate contraception (as defined below) from the first day of Screening prior to study entry, for the duration of study participation and for at least 120 days following their last study treatment day.

c. Adequate contraception includes sexual abstinence (only if preferred method of birth control); oral, intravaginal or transdermal combined estrogen and progesterone hormonal contraception associated with inhibition of ovulation; oral, injectable or implantable progesterone-only hormonal contraception associated with inhibition of ovulation; intrauterine device (IUD); intrauterine hormone-releasing system (IUS); bilateral tubal occlusion; or only vasectomized sexual partner(s).

Exclusion Criteria:

A patient will be excluded from study participation if ANY of the following criteria apply:

1. Patients who are planning to receive intratumoural treatment or radiotherapy to any of the intended target tumours within 4 weeks prior to Screening, or during treatment with tigilanol tiglate or pembrolizumab, or who have received radiotherapy within 2 weeks of the start of study treatment. (Note: Patients must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 4-week washout is permitted for palliative radiation [≤4 weeks of radiotherapy] to non-CNS disease).
2. A tumour intended for injection that is immediately adjacent to, or with infiltration into, any major artery or vein.
3. A tumour intended for injection located in an area where post-injection swelling could compromise the airway.
4. Any previous intervention in the area of the intended injected tumour in proximity of the airway (such that tracking of the injected fluid may be unpredictable and could lead to airway swelling).
5. A histologically confirmed diagnosis of uveal or mucosal melanoma as the only intended injected tumour.
6. Have a positive urine pregnancy test within 72 hours prior to start of study treatment (Note: If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required).
7. Have received a live vaccine within 30 days prior to the start of study treatment. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG) and typhoid vaccine. (Note: Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines [e.g., FluMist®] are live attenuated vaccines and are not allowed).
8. Are planning to receive concomitant other biologic therapy, hormonal therapy, other chemotherapy to treat their melanoma while on study treatment.
9. Have received any of the following within 4 weeks prior to the start of study treatment; systemic anticancer therapy, including investigational agents, or has participated in a study of an investigational agent or has used an investigational device. (Note: Patients who have entered the follow-up phase of an investigational study may participate as long as it has been at least 4 weeks after the last dose of the previous investigational agent). Patients must have recovered from all AEs due to previous therapies to ≤ Grade 1 or baseline patients with ≤ Grade 2 neuropathy may be eligible. (Note: If patient received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting study treatment). (Note: Patients who have received systemic anticancer therapy can be considered for inclusion provided a washout period of 4 weeks or 5 half-lives, whichever is shorter, has occurred).
10. Have known, current or history of central nervous system metastases, active cerebral metastasis and/or carcinomatous meningitis.
11. Have any bleeding diathesis or coagulopathy, or are taking warfarin, that would make intratumoural injection or biopsy unsafe.
12. Clinically significant acute or unstable cardiovascular, cerebrovascular disorders.
13. Patients with significant peripheral vascular disease whose accessible tumours intended for injection are located in their extremities.
14. Have prior allogeneic tissue/solid organ transplant.
15. Have a history of allergic reactions or severe hypersensitivity (Grade ≥ 3) attributed to tigilanol tiglate or pembrolizumab, compounds of similar chemical or biologic composition to tigilanol tiglate or pembrolizumab, any of their excipients or other agents used in the study, or have experienced unacceptable toxicity to a checkpoint inhibitor.
16. Have an active infection requiring systemic therapy.
17. Have known immunodeficiency or are receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the start of study treatment.
18. Have a known additional malignancy that is progressing or has required active treatment within the past 3 years. (Note: Patients with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ [e.g., breast carcinoma, or cervical cancer in situ] that have undergone potentially curative therapy are not excluded).
19. Have active autoimmune disease that has required systemic treatment in the past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs). (Note: Replacement therapy [e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency] is not considered a form of systemic autoimmune treatment and is allowed).
20. Have a history of non-infectious pneumonitis / interstitial lung disease that required steroids or has current pneumonitis / interstitial lung disease.
21. Have known human immunodeficiency virus (HIV) and/or history of Hepatitis B or Hepatitis C viral infections, or known to be positive for Hepatitis B antigen (HbsAg), Hepatitis B virus (HBV) DNA or Hepatitis C Antibody or RNA. (Note: Active Hepatitis C virus [HCV] is defined by a known positive Hepatitis C Antibody result and known quantitative HCV RNA results greater than the lower limits of detection of the assay).
22. Have a known psychiatric or substance abuse disorder that would interfere with the patient's ability to cooperate with the requirements of the study.
23. Have a history of or current evidence of any condition, therapy or laboratory abnormality that might confound the results of the study, interfere with the patient's participation for the full duration of the study, or is not in the best interest of the patient to participate, in the opinion of the treating Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2021-05-07 (Actual); Primary Completion 2022-07-12 (Actual); Study Completion 2022-07-12 (Actual)

PRIMARY OUTCOMES:
Determine Dose Level | 12 months
  To determine the dose level of intratumoural tigilanol tiglate when administered in combination with pembrolizumab (200 mg IV) at which there is no dose-limiting toxicity (DLT) recorded.
Determine incidence of Treatment Emergent Adverse Events | 12 months
  To determine the incidence of Treatment Emergent Adverse Events (TEAEs) including all grades of TEAEs and abnormal laboratory finding AEs

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | 24 months
  To assess the Objective Response Rate (ORR) includes partial response (PR) and complete response (CR) of injected tumours as well as non-injected tumours.
Best Overall Response (BOR) | 24 months
  To assess the Best Overall Response (BOR) of injected as well as non-injected tumours.
Durable Response Rate (DRR) | 24 months
  To assess the Durable Response Rate (DRR) of injected tumours.
Duration of Response (DoR) | 24 months
  To assess the Duration of Response (DoR) of injected tumours
Progression Free Survival (PFS) | 24 months
  To assess the Progression Free Survival (PFS). Defined as the length of time during and after treatment that a patient lives without disease progression.
Incidence of treatment related and non-treatment related Treatment Emergent Adverse Events (TEAEs) and abnormal laboratory tests. | 24 months
  All Grade ≥ 3 TEAEs, serious (including fatal) AEs (SAEs), and TEAEs defined as events of interest by the Investigator.
  Grading will be as per 'Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0, 2017'. The CTCAE scale is measured from Grade 1 (mild) to Grade 5 (death).

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Georgina Long, BSc PhD MBBS FRACP FAHMS, Principal Investigator — Melanoma Institute Australia; Dr Megan Lyle, BMed FRACP, Principal Investigator — Cairns and Hinterland Hospital and Health Service; Dr Melvin Chin, Principal Investigator — Prince of Wales Hospital
Locations (2):
- Australia (2):
  - Melanoma Institute Australia, Wollstonecraft, New South Wales
  - Cairns and Hinterland Hospital and Health Service, Cairns, Queensland